CLINICAL TRIAL: NCT07309497
Title: Pragmatic Geriatric Assessment (pGA) Before Bispecific Antibody and CAR-T-Cell Therapy (GA-ACT Trial) for the Prediction of Toxicity and Outcomes in Older Patients Scheduled for Chimeric Antigen Receptor T-Cell Therapy (CAR-T-Cell-Therapy) or Bispecific Antibody (bsAB) Treatment
Brief Title: Pragmatic Geriatric Assessment Before CAR-T or Bispecific Antibody Therapy to Predict Side Effects and Outcomes in Older Patients (GA-ACT Trial)
Acronym: GA-ACT
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other); Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC-No 2025-01228; KLS-6127-08-2024-R (Other Grant/Funding Number: Krebsliga Schweiz)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma (MM), Lymphoma, Large B-Cell, Diffuse (DLBCL), Lymphoma; CART Therapy; Bispecific Antibody; Geriatric Hematology
Keywords: geriatric assessment; lymphoma; multiple myeloma; bispecific antibodies; chimeric antigen receptor; outcome assessment; toxicity; health related quality of life
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- geriatric assessment group
  Interventions: Other: pragmatic geriatric assessment

INTERVENTIONS:
Other: pragmatic geriatric assessment — observational study
Other: pragmatic geriatric assessment — pragmatic geriatric assessment

SUMMARY:
CAR-T cell or bispecific antibody therapies are a new treatment option for adult patients with aggressive forms of lymphoma or so-called plasma cell diseases ('multiple myeloma', 'plasma cell myeloma') that could not be cured with other, less intensive approaches. However, these are intensive therapies that can be associated with severe and potentially life-threatening side effects. Although there is no age limit for these therapies, we know little about the short- and long-term side effects of these treatments in people of advanced age.

Although a small number of patients in the pivotal studies were even over 80 years old, their number was too small to be able to assess the tolerability and success specifically in people over 65. At present, the treating physicians decide whether and, if so, which patients are considered 'fit' enough for this therapy. An objective assessment of the kind we want to investigate in our study does not currently exist on a regular basis. In this study, we therefore want to use simple clinical methods to investigate the effects of these forms of therapy in different areas of everyday function that are important for people in older age (mobility, memory, self-care skills, nutrition). We want to find out whether these investigations help to predict the risk of severe and/or long-term side effects. Based on the results, a pragmatic geriatric assessment could be introduced as standard before these therapies. Older patients could thus expect an improvement in their quality of life thanks to more predictable risks and side effects. Standardized screening could lead to lower healthcare costs for treatment and aftercare for both forms of therapy.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients age ≥ 65 years,
* scheduled for CAR-T-cell or bsAB treatments
* signed informed consent
* sufficient knowledge of the German or French language

Exclusion Criteria:

* inability to understand or sign informed consent
* refuse to consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients age ≥ 65 years and older, treated at the University Hospitals in Bern and Zurich and undergoing CAR-T-cell or bsAB therapy
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
treatment toxicity | From enrollment to 3 month after end of treatment
  primary endpoint will be the composite rate of death or any one of ≥ grade 3 toxicity

SECONDARY OUTCOMES:
health related quality of life | From enrollment to 3 month after end of treatment
  Secondary endpoints will be the rate of transfer to intensive care units, the length of hospital stay, the discharge home versus to rehab or nursing-care facilities as well as changes in physical function, cognitive function, nutritional status, ability of self-care and the quality-of-life at discharge and three months after start of therapy. In addition premature CAR-T or bsAB discontinuation, the frequency of treatment-specific toxicities such as the cytokine-release syndrome (CRS) and the immune effector cell-associated neurotoxicity syndrome (ICANS) will be captured

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke Rösler, Dr. med., Principal Investigator — Universitätsspital Zürich
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
under discussion